CLINICAL TRIAL: NCT02392871
Title: An Open-label, Single-arm, Phase I/II, Multicentre Study to Evaluate the Safety and Efficacy of the Combination of Dabrafenib, Trametinib and Palliative Radiotherapy in Patients with Unresectable (stage IIIc) and Metastatic (stage IV) BRAF V600E/K Mutation-positive Cutaneous Melanoma
Brief Title: Radiotherapy & Combi in Metastatic Melanoma
Acronym: CombiRT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Collaborators: Melanoma Institute Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02.14
Record Dates: First submitted 2015-03-10; First posted 2015-03-19 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic melanoma; Palliative radiotherapy
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy (Experimental): Palliative radiotherapy in combination with dabrafenib and trametinib Eligible subjects are patients who have been on dabrafenib and trametinib for more than 2 weeks, as the current standard management for advanced stage melanoma.
  Palliative RT will be delivered to symptomatic or bulky (>2cm) soft tissue, nodal or bony metastases concurrently with dabrafenib and trametinib. Up to 3 areas of disease can be irradiated at the same time.
  Following RT, dabrafenib and trametinib alone will be continued until disease progression according to RECIST 1.1 criteria.
  Interventions: Radiation: Palliative radiotherapy; Drug: Dabrafenib and trametinib (combination)

INTERVENTIONS:
Radiation: Palliative radiotherapy
Drug: Dabrafenib and trametinib (combination) — Patients should be taking dabrafenib and trametinib for at least 2 weeks prior to enrolment into the study.

SUMMARY:
The purpose of this study is to investigate the side effects and safety, and effectiveness of combining dabrafenib and trametinib with radiotherapy.

Previous and ongoing clinical trials have demonstrated the effectiveness and safety of combining both dabrafenib and trametinib compared with dabrafenib alone. This has led to the approval for the use of both drugs in combination in people with metastatic melanoma with the BRAF mutation. Melanoma that has spread to other parts of the body may also benefit from radiotherapy to help reduce symptoms from melanoma. Previous studies have shown that melanoma may be sensitive to radiotherapy and that it can help to improve quality of life.

The intention of the CombiRT study is to establish if dabrafenib, trametinib and radiotherapy combined is a safe and effective treatment for metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. Signed written informed consent.
3. Histologically confirmed cutaneous melanoma that is either Stage IIIC (unresectable) or Stage IV (metastatic), and determined to be BRAF V600E/K mutation-positive as determined by a BRAF mutation assay.

   Note: For Stage IIIC disease, the decision that the disease is unresectable should be formally endorsed by the melanoma multidisciplinary tumour board of the local institution.
4. Have received dabrafenib and trametinib for 2 weeks or more prior to enrolment in the study (i.e. first fraction of palliative RT), and is still continuing with dabrafenib and trametinib.
5. Symptomatic or bulky (greater than 2 cm in diameter) soft tissue, nodal or bony metastases requiring palliative RT.
6. Have measurable disease according to RECIST 1.1 criteria. Note: patients with bony metastases that are not measurable by RECIST 1.1 criteria are allowed in this study.
7. All anti-cancer treatment-related toxicities (except alopecia and laboratory values as listed on Table 1 in protocol) must be less than or equal to (≤) Grade 1 according to the Common Terminology Criteria for Adverse Events version 4 (CTCAE version 4.03; NCI, 2009) at the time of study enrolment.
8. Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
9. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrolment and agree to use effective contraception, from 14 days prior to enrolment throughout the treatment period, and for 4 months after the last dose of study treatment.
10. An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
11. Adequate baseline organ function (as defined in Table 1 in protocol).

Exclusion Criteria:

1. Treatment with Ipilimumab or any other anti-CTLA-4 monoclonal antibody therapy within the past 4 weeks.
2. Treatment with anti-PD-1 or anti-PD-L1 monoclonal antibody therapy within the past 4 weeks.
3. Known ocular or primary mucosal melanoma.
4. Four (4) or more lesions requiring palliative RT at the time of study enrolment.
5. Symptomatic brain metastases or those treated < 3 months previously.
6. Clear evidence of systemic disease progression on dabrafenib and trametinib.
7. Systemic anti-cancer treatment (chemotherapy, immunotherapy, biologic therapy, vaccine therapy, or investigational treatment) within the last 4 weeks. Prior interferon treatment in the adjuvant setting is allowed.

   Note: Tamoxifen and aromatase inhibitors are allowed in the adjuvant setting of breast cancer.
8. Current use of a prohibited medication (list of prohibited medications in protocol).
9. History of malignancy other than disease under study within 3 years of study enrolment with exceptions below, or any malignancy with confirmed activating RAS mutation.

   Note: Prospective RAS testing is not required. However, if the results of previous RAS testing are known, they must be used in assessing eligibility.

   Exception: Subjects who have been disease-free for 3 years, or subjects with a history of completely resected non-melanoma skin cancer.
10. Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures.
11. A history of known Human Immunodeficiency Virus (HIV).
12. A history or evidence of cardiovascular risk including any of the following:

    * A QT interval corrected for heart rate using the Bazett's formula (QTcB) ≥ 480 msec;
    * A history or evidence of current clinically significant uncontrolled arrhythmias;
    * A history of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within 6 months prior to enrolment;
    * A history or evidence of current ≥ Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines;
    * Patients with intra-cardiac defibrillators;
    * Abnormal cardiac valve morphology (≥ grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study; g. Treatment refractory hypertension defined as a blood pressure of systolic> 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy; h. Known cardiac metastases.
13. A history of retinal vein occlusion (RVO).
14. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO).
15. Pregnant or nursing females.
16. Previous RT to the same lesion or area due to receive the current course of palliative RT.

    Note: patients who had previous RT to other areas are eligible to the study if the previous RT was completed more than 8 weeks prior.
17. A history of autoimmune diseases which are known to increase radiation toxicity, including systemic lupus erythematosus and scleroderma.
18. Genetic syndromes exhibiting increased radiosensitivity (e.g. ataxia telangiectasia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Toxicity profile for patients receiving dabrafenib and trametinib in combination with RT, by measuring adverse events and radiotherapy associated toxicities. | 0-12 months

SECONDARY OUTCOMES:
Patients' pain using a visual analog scale (questionnaire) | 0-12 months
Overall disease response by measuring progression free survival and overall survival. | 0-12 months
Local treatment response in the irradiated index lesion(s). | 0-12 months
Time to local progression in the irradiated index lesion(s). | 0-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tim Wang, Principal Investigator — Westmead Hospital
Locations (3):
- Australia (3):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: No